CLINICAL TRIAL: NCT06843044
Title: An Open-label, Comparative, Randomized, Multicenter Phase IV Clinical Study to Evaluate the Clinical Efficacy and Safety of the Drug Ranquilon, Tablets, 1 mg, in Patients With Anxiety Disorders Due to Neurasthenia and Adjustment Disorders
Brief Title: Efficacy and Safety of Ranquilon in Patients With Anxiety Disorders Due to Neurasthenia and Adjustment Disorders
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAN-04-05-2024
Record Dates: First submitted 2025-02-17; First posted 2025-02-24 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Neurasthenia; Adjustment Disorders
MeSH Terms: conditions — Anxiety Disorders; Neurasthenia; Adjustment Disorders | interventions — GB-115; 2-((2-morpholino)ethylthio)-5-ethoxybenzimidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranquilon, 6 mg/day (Experimental): Ranquilon, 1 mg tablets, at a dosage of 6 mg/day for 28 days
  Interventions: Drug: Ranquilon
- Afobazole, 30 mg/day (Active Comparator): Afobazole, 10 mg tablets, at a dosage of 30 mg/day for 28 days
  Interventions: Drug: Afobazole

INTERVENTIONS:
Drug: Ranquilon — 1 mg tablets
  Other Names: GB-115; N-(6-phenylhexanoyl)glycyl-L-tryptophan amide
  Arms: Ranquilon, 6 mg/day
Drug: Afobazole — 10 mg tablets
  Other Names: Fabomotizole
  Arms: Afobazole, 30 mg/day

SUMMARY:
Study is to evaluate the efficacy and safety of the drug Ranquilon, 1 mg tablets, at a dosage of 6 mg/day compared to the drug Afobazole, 10 mg tablets, at a dosage of 30 mg/day for the treatment of patients with anxiety disorders due to neurasthenia and adjustment disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 to 70 years;
2. Written informed consent form in accordance with current legislation;
3. Patients with anxiety and established diagnoses based on ICD-10 criteria: neurasthenia (F48.0) or adjustment disorder (F43.2);
4. Anxiety severity on the HARS scale of 18-24 points;
5. Assessment of the severity of suicidal thoughts using the Columbia scale <3 points;
6. Severity of asthenia on the Multidimensional Fatigue Inventory Scale (MFI-20) greater than 50 points;
7. Total score on the Hamilton Depression Rating Scale (HAMD-17) < 6;
8. Score on the CGI-s scale of at least 4 points;
9. Negative pregnancy test for women of childbearing potential;
10. Agreement to use effective contraceptive methods throughout the study and for 30 days after its completion (for women of childbearing potential and men);
11. Ability to understand the requirements of the study, provide written informed consent (including consent for the use and disclosure of health-related information), and comply with the procedures outlined in the study protocol.

Non-inclusion Criteria:

1. Known intolerance to the active and/or excipient substances contained in the study drugs;
2. Known lactase deficiency, lactose intolerance, glucose-galactose malabsorption, or galactose intolerance;
3. Patients requiring prohibited concomitant therapy within this study (MAO inhibitors, antidepressants, neuroleptics, anxiolytics and sedatives (including herbal), hypnotics when used on a regular basis), or who have taken these medications within the last month;
4. Established or suspected alcohol/narcotic substance use at the time of screening or randomization, and/or a history of alcohol, narcotic, or drug dependence;
5. Presence of oncological diseases, including in history (except for cured tumors with stable remission for more than 5 years);
6. Tuberculosis, including in history;
7. Presence of HIV, chronic viral hepatitis B/C, syphilis (including past history), or a positive test for HIV, hepatitis B/C, or syphilis at screening;
8. Patients with a diagnosis of other anxiety disorders (F41) established based on ICD-10 criteria;
9. Schizophrenia, schizoaffective disorders, affective disorders, and panic disorders;
10. Acute psychosis (endogenous-processual, organic, or somatogenic), including in history;
11. Organic lesions of the central nervous system of traumatic and alcoholic origin;
12. Post-encephalitic syndrome;
13. History of brain tumors (including past diagnoses);
14. Degenerative diseases of the central nervous system (CNS), particularly multiple sclerosis;
15. History of depression (including past episodes);
16. Suicide attempts in history;
17. Generalized anxiety disorder, including in history;
18. History of epilepsy and seizures (including past episodes);
19. Decompensated diabetes mellitus;
20. Established diagnosis of chronic kidney disease stage 3A and above, or estimated glomerular filtration rate (eGFR) calculated by the Cockcroft-Gault formula ≤ 59 ml/min/1.73 m²;
21. Established diagnosis of liver failure of any severity, or elevated levels of ALT, AST or total bilirubin >3 times the upper limit of normal according to laboratory standards;
22. History of major surgical interventions within six months prior to screening;
23. Chronic heart failure III-IV functional class according to the New York Heart Association (NYHA) classification;
24. Severe, decompensated, or unstable diseases (any diseases or conditions that poses a life-threatening risk to the patient, worsens the patient's prognosis, or makes participation in the clinical study impossible);
25. Pregnant women, breastfeeding women, or women planning to become pregnant during the study or within 30 days after participation ends;
26. Refusal by the patient to use permitted methods of contraception or to completely abstain from sexual contact throughout the entire period of participation in the study starting from Visit 0 and for 30 days after completion of participation;
27. Current participation or planned participation by the patient in psychological or psychotherapeutic activities aimed at treating anxiety disorder during the clinical trial period;
28. Participation in any other clinical trial within 90 days prior to the start of the screening period;
29. Lack of patient cooperation;
30. Other reasons, at the investigator's discretion, that may hinder the patient's participation in the study or pose unjustified risk to the patient.

Exclusion Criteria:

1. The patient's decision to withdraw from the study (revocation of informed consent);
2. Each patient has the right to discontinue participation in the study at any time without explanation. Withdrawal from the study will not affect the medical care provided to the patient in the future;
3. The investigator's decision that the patient needs to be excluded in the best interest of the patient;
4. The patient refuses to cooperate with the investigator or is non-compliant;
5. Emergence of reasons/situations during the study that threaten the patient's safety (e.g., hypersensitivity reactions, serious adverse events, etc.);
6. Inclusion of a patient in the study that does not meet the inclusion/exclusion criteria, including cases of deviation from normal values in laboratory test results obtained at Visit 0;
7. Significant violation of the treatment regimen.

   A significant violation is considered:
   1. Missing doses of the study drugs for 2 consecutive days or more, or
   2. Taking a total number of tablets < 80% or > 120% of the full course (the full course for Ranquilon is 168 tablets, and for Afobazole, it is 84 tablets).
8. Positive pregnancy test;
9. Confirmed diagnosis of COVID-19;
10. Emergence of other reasons during the study that prevent its conduct according to the protocol;
11. Patient death;
12. Sponsor-initiated study termination;
13. Termination of the study by the Investigator;
14. Termination of the study by regulatory authorities.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a significant reduction in anxiety levels (by 50% or more) on Hamilton Anxiety Rating Scale (HARS) compared to baseline on Day 29 ± 1 (Visit 3) | Day 29 ± 1 (Visit 3)
  HARS scale includes 14 items, each of which is rated on the Likken scale (from 0 points as absence of the symptom to 4 points as the worst possible symptom). Of these, 13 items relate to the manifestation of anxiety in daily life, 14th item relate to the manifestation of anxiety during examinations.

SECONDARY OUTCOMES:
Change in anxiety levels according to the Hamilton Anxiety Rating Scale (HARS) scale on Day 29 ± 1 (Visit 3) compared to baseline | Day 29 ± 1 (Visit 3)
  HARS scale includes 14 items, each of which is rated on the Likken scale (from 0 points as absence of the symptom to 4 points as the worst possible symptom). Of these, 13 items relate to the manifestation of anxiety in daily life, 14th item relate to the manifestation of anxiety during examinations.
Proportion of patients with a reduction in anxiety levels on the Hamilton Anxiety Rating Scale (HARS) scale to 17 points or less on Day 29 ± 1 (Visit 3) | Day 29 ± 1 (Visit 3)
  HARS scale includes 14 items, each of which is rated on the Likken scale (from 0 points as absence of the symptom to 4 points as the worst possible symptom). Of these, 13 items relate to the manifestation of anxiety in daily life, 14th item relate to the manifestation of anxiety during examinations.
Proportion of patients with a score of 2 points or less on the Clinical Global Impression (CGI-s) scale as assessed by the physician (healthy or borderline disorder) on Day 29 ± 1 (Visit 3) | Day 29 ± 1 (Visit 3)
  The scale ranges from 1 to 7 points, where 1 indicates healthy and 7 indicates very severe disorder.
Change in the severity of the patient's condition on the Clinical Global Impression (CGI-s) scale by Day 29 ± 1 (Visit 3) compared to baseline | Day 29 ± 1 (Visit 3)
  The scale ranges from 1 to 7 points, where 1 indicates healthy and 7 indicates very severe disorder.
Change in the total score on the Multidimensional Fatigue Inventory (MFI-20) on Day 29 ± 1 (Visit 3) compared to baseline | Day 29 ± 1 (Visit 3)
  If the total score on any of the subscales (General Fatigue, Reduced Activity, Decreased Motivation, Physical Fatigue, Mental Fatigue) is above 12, it may serve as preliminary grounds for diagnosing "asthenic syndrome." Each subscale is assessed from 4 points (lack of symptoms) to 20 points (worst symptoms possible).
Proportion of patients with a reduction in total score on the Multidimensional Fatigue Inventory (MFI-20) by 25% on Day 29 ± 1 (Visit 3) compared to baseline | Day 29 ± 1 (Visit 3)
  Normally, the total number of points should not exceed 30. If the total score on any of the subscales (General Fatigue, Reduced Activity, Decreased Motivation, Physical Fatigue, Mental Fatigue) is above 12, it may serve as preliminary grounds for diagnosing "asthenic syndrome." Each subscale is assessed from 4 points (lack of symptoms) to 20 points (worst symptoms possible).
Proportion of patients with a reduction in total score on the Multidimensional Fatigue Inventory (MFI-20) by 50% on Day 29 ± 1 (Visit 3) compared to baseline | Day 29 ± 1 (Visit 3)
  Normally, the total number of points should not exceed 30. If the total score on any of the subscales (General Fatigue, Reduced Activity, Decreased Motivation, Physical Fatigue, Mental Fatigue) is above 12, it may serve as preliminary grounds for diagnosing "asthenic syndrome." Each subscale is assessed from 4 points (lack of symptoms) to 20 points (worst symptoms possible).
Proportion of patients with a total score on the Multidimensional Fatigue Inventory (MFI-20) reduced to 30 points or less on Day 29 ± 1 (Visit 3) | Day 29 ± 1 (Visit 3)
  Normally, the total number of points should not exceed 30. If the total score on any of the subscales (General Fatigue, Reduced Activity, Decreased Motivation, Physical Fatigue, Mental Fatigue) is above 12, it may serve as preliminary grounds for diagnosing "asthenic syndrome." Each subscale is assessed from 4 points (lack of symptoms) to 20 points (worst symptoms possible).
Absolute value of the patient's self-assessment of their subjective condition for all individual items on the Multidimensional Fatigue Inventory (MFI-20) scale by Day 29 ± 1 (Visit 3) | Day 29 ± 1 (Visit 3)
  Normally, the total number of points should not exceed 30. If the total score on any of the subscales (General Fatigue, Reduced Activity, Decreased Motivation, Physical Fatigue, Mental Fatigue) is above 12, it may serve as preliminary grounds for diagnosing "asthenic syndrome." Each subscale is assessed from 4 points (lack of symptoms) to 20 points (worst symptoms possible).
Change in total score on the Columbia-Suicide Severity Rating Scale (C-SSRS) by Day 29 ± 1 (Visit 3) compared to baseline | Day 29 ± 1 (Visit 3)
  A severity rating of "3" or higher indicates a serious risk of suicide. A rating of "5" and any identified suicidal actions indicate an extremely high risk and an absolute necessity for urgent therapeutic measures and hospitalization. The section "intensity of suicidal thoughts" allows for a more accurate assessment of severity and prediction of its dynamics.
Change in total score on the Emotional Eating Questionnaire by Day 29 ± 1 (Visit 3) compared to baseline | Day 29 ± 1 (Visit 3)
  The scale ranges from 0 to 30 points, where a minimum indicates no emotional overeating and a maximum indicates a strong dependence of eating behavior on emotional state.
Change in total score on the Psychological Stress Measure (PSM-25) by Day 29 ± 1 (Visit 3) compared to baseline | Day 29 ± 1 (Visit 3)
  A score below 99 indicates low stress, a score between 100-125 indicates moderate stress; a score above 125 indicates high stress
Safety and Tolerability: adverse event (AE) rate | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 43 ± 1 for each participant
  Number and frequency of adverse events (AEs) or serious AEs (SAEs)
Safety and Tolerability: AEs associated with the study drug | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 43 ± 1 for each participant
  Number and frequency of AEs or SAEs associated with the study drug
Safety and Tolerability: treatment discontinuation | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 43 ± 1 for each participant
  Percentage of patients who discontinued treatment due to the occurrence of AEs/SAEs
Safety and Tolerability: vital signs - systolic blood pressure (SBP) | Screening, day 1, day 29 ± 1, day 43 ± 1
  SBP, mmHg
Safety and Tolerability: vital signs - diastolic blood pressure (DBP) | Screening, day 1, day 29 ± 1, day 43 ± 1
  DBP, mmHg
Safety and Tolerability: vital signs - respiratory rate (RR) | Screening, day 1, day 29 ± 1, day 43 ± 1
  RR, breaths per minute
Safety and Tolerability: vital signs - heart rate (HR) | Screening, day 1, day 29 ± 1, day 43 ± 1
  HR, beats per minute
Safety and Tolerability: vital signs - body temperature | Screening, day 1, day 29 ± 1, day 43 ± 1
  Body temperature, Celsius scale
Safety and Tolerability: concomitant treatment | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 43 ± 1 for each participant
  Data on concomitant treatment (if any)
Safety and Tolerability: clinical blood test - hemoglobin | Screening, day 29 ± 1
  Hemoglobin (g/L)
Safety and Tolerability: clinical blood test - hematocrit | Screening, day 29 ± 1
  Hematocrit (%)
Safety and Tolerability: clinical blood test - red blood cell count | Screening, day 29 ± 1
  Red blood cell count (cells/L)
Safety and Tolerability: clinical blood test - platelet count | Screening, day 29 ± 1
  Platelet count (cells/L)
Safety and Tolerability: clinical blood test - leukocyte count | Screening, day 29 ± 1
  Leukocyte count (cells/L)
Safety and Tolerability: clinical blood test - erythrocyte sedimentation rate | Screening, day 29 ± 1
  Erythrocyte sedimentation rate (mm/h)
Safety and Tolerability: clinical blood test - myelocytes | Screening, day 29 ± 1
  Leukocyte formula (myelocytes, %)
Safety and Tolerability: clinical blood test - band neutrophils | Screening, day 29 ± 1
  Leukocyte formula (band neutrophils, %)
Safety and Tolerability: clinical blood test - segmented neutrophils | Screening, day 29 ± 1
  Leukocyte formula (eosinophils, %)
Safety and Tolerability: clinical blood test - basophils | Screening, day 29 ± 1
  Leukocyte formula (basophils, %)
Safety and Tolerability: clinical blood test - monocytes | Screening, day 29 ± 1
  Leukocyte formula (monocytes, %)
Safety and Tolerability: clinical blood test - lymphocytes | Screening, day 29 ± 1
  Leukocyte formula (lymphocytes, %)
Safety and Tolerability: urinalysis - specific gravity | Screening, day 29 ± 1
  Specific gravity of the urine
Safety and Tolerability: urinalysis - color | Screening, day 29 ± 1
  Color of the urine
Safety and Tolerability: urinalysis - transparency | Screening, day 29 ± 1
  Transparency of the urine
Safety and Tolerability: urinalysis - pH | Screening, day 29 ± 1
  pH of the urine
Safety and Tolerability: urinalysis - protein | Screening, day 29 ± 1
  Protein concentration (g/L)
Safety and Tolerability: urinalysis - glucose | Screening, day 29 ± 1
  Glucose concentration (mmol/L)
Safety and Tolerability: urinalysis - red blood cells | Screening, day 29 ± 1
  Red blood cell content (number in sight)
Safety and Tolerability: urinalysis - white blood cells | Screening, day 29 ± 1
  White blood cell content (number in sight)
Safety and Tolerability: urinalysis - epithelial cells | Screening, day 29 ± 1
  Epithelial cell content (number in sight)
Safety and Tolerability: urinalysis - ketone bodies | Screening, day 29 ± 1
  Ketone bodies (mmol/L)
Safety and Tolerability: urinalysis - urobilinogen | Screening, day 29 ± 1
  Urobilinogen (mcmol/L)
Safety and Tolerability: blood chemistry - glucose | Screening, day 29 ± 1
  Glucose concentration (mmol/L)
Safety and Tolerability: blood chemistry - cholesterol | Screening, day 29 ± 1
  Total cholesterol concentration (mmol/L)
Safety and Tolerability: blood chemistry - protein | Screening, day 29 ± 1
  Total protein concentration (g/L)
Safety and Tolerability: blood chemistry - bilirubin | Screening, day 29 ± 1
  Total bilirubin concentration (micromol/L)
Safety and Tolerability: blood chemistry - creatinine | Screening, day 29 ± 1
  Creatinine concentration (micromol/L)
Safety and Tolerability: blood chemistry - alkaline phosphatase | Screening, day 29 ± 1
  Alkaline phosphatase activity (U/L)
Safety and Tolerability: blood chemistry - alanine transaminase | Screening, day 29 ± 1
  Alanine transaminase activity (U/L)
Safety and Tolerability: blood chemistry - aspartate transaminase | Screening, day 29 ± 1
  Aspartate transaminase activity (U/L)
Safety and Tolerability: blood chemistry - urea | Screening, day 29 ± 1
  Urea concentration (mmol/L)

CONTACTS AND LOCATIONS:
Locations (6):
- Russia (6):
  - Engels Psychiatric Hospital State Health Care Institution of the Ministry of Health of the Saratov Region, Engel's
  - Unimed-C Jsc, Moscow
  - Aurora MedFort LLC, Saint Petersburg
  - Limited Liability Company "Research Center Eco-Safety", Saint Petersburg
  - Limited Liability Company "Stepmed Clinic", Saint Petersburg
  - Saratov City Psychoneurological Dispensary, Saratov

IPD SHARING:
Plan to Share IPD: No